CLINICAL TRIAL: NCT02438904
Title: Compassionate Access of the Miltenyi Device for CD34+ Cell Selection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-0295; NCI-2015-00979 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Blood And Marrow Transplantation
Keywords: Blood And Marrow Transplantation; Stem cell transplantation; SCT; Poor graft function; CD34+ cell infusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- CD34 Positive Stem Cell Infusion (Experimental): Participants infused by vein with around 1 - 4 million/kg CD34+ selected cells. If the first infusion is not effective, an additional infusion may be given 4 - 6 weeks after the first infusion.
  Interventions: Biological: CD34 Positive Stem Cell Infusion; Device: Miltenyi device

INTERVENTIONS:
Biological: CD34 Positive Stem Cell Infusion — Participants infused by vein with around 1 - 4 million/kg CD34+ selected cells.
Device: Miltenyi device — Miltenyi device is used for CD34+ cell infusions) to patients who experience poor graft function after stem cell transplantation (SCT).
  Other Names: CliniMACS device

SUMMARY:
Objectives:

Primary Objective

To provide compassionate access to the Miltenyi device for CD34+ cell infusions to patients who experience poor graft function after stem cell transplantation (SCT).

DETAILED DESCRIPTION:
The therapy that you will receive involves you being given an infusion of CD34 positive stem cells.

Below is a detailed explanation of the therapeutic procedures that will be performed.

CD34 positive stem cells infusion:

The CD34 positive stem cells are collected from a donor's blood. The blood cells go through CD34 (stem cell) selection process that collects the stem cells that are needed for the infusion. This process collects the early immune cells your body will need to regrow your immune system, and makes sure that other cells will not be infused. This process will decrease (but not eliminate completely) the other types of cells. If you agree to receive this treatment, the CD34 cells will then be infused into your body.

The CD34 positive cells will be given by vein in either an inpatient or outpatient treatment area. The infusion will last about 10-30 minutes.

Before the infusion, you will receive Tylenol (acetaminophen) by mouth and Benadryl (diphenhydramine hydrochloride) by mouth or vein about 30-60 minutes before the infusion. These drugs will be used to help lower the risk of side effects. If side effects occur during the infusion, the doses of the drugs may be adjusted (up or down) until the symptoms are gone. Also, if you have side effects during the infusion, you will be observed for 2 hours after it is given or until the symptoms have stopped completely (whichever is later). During this time, your blood pressure, heart rate, breathing rate, temperature, and the level of oxygen in your blood will be checked every 15-30 minutes.

About 4-6 weeks after the first infusion, you may receive an additional infusion, if your doctor thinks it is needed.

Clinic Visits:

One (1) time a week after the infusion, until your doctor thinks it is no longer clinically needed, you will have the following tests:

* Blood (about 1 teaspoon) will be drawn for routine tests.
* You will be checked for signs of graft versus host disease (GVHD). Symptoms of GVHD include skin rash, nausea, vomiting, diarrhea, and abnormal liver function.

This is an investigational study. The CD34 positive stem cell infusion to help boost cell counts is not FDA approved.

Up to 75 patients will be enrolled on this treatment.

ELIGIBILITY:
Inclusion Criteria:

1) Patients who have poor or no graft function post stem cell transplantation.

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-05-06 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Increased Graft Function after Stem Cell Transplantation (SCT) | 4 weeks
  Blood drawn for signs of graft versus host disease (GVHD).

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Shpall, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/04/NCT02438904/ICF_000.pdf